CLINICAL TRIAL: NCT04844463
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-68179280 in Healthy Participants
Brief Title: A Study of JNJ-68179280 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108989; 68179280IBD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive a single ascending oral dose of JNJ-68179280 or placebo capsules under fasted condition (Cohort 1, 2 and 5) and under fasted-fed condition (either Cohort 3 or 4) on Day 1. In 1 of the study cohorts 3 or 4, participants will also receive study intervention on Day 8 under fed condition. One additional optional Cohort 6 may be dosed to assess the safety and pharmacokinetics (PK) of an alternate dose of formulation A under fasted condition.
  Interventions: Drug: JNJ-68179280; Other: Placebo
- Part 2: Multiple Ascending Dose (MAD) (Experimental): Participants will receive multiple ascending oral doses of JNJ-68179280 or placebo capsules once daily in Cohort 1 through 4 or twice daily in Cohort 5 (optional) on Days 1 through 14 under fasted or fed condition.
  Interventions: Drug: JNJ-68179280; Other: Placebo
- Part 3: Multiple Dose Alternative Formulation (Optional) (Experimental): Participants will receive multiple oral doses of an alternative JNJ-68179280 formulation once daily in Cohort 1 and Cohort 2 (optional) on Days 1 through 14 under fasted or fed condition. Doses in Part 3 will depend on the safety, tolerability, PK and pharmacodynamics data from Part 1 and Part 2.
  Interventions: Drug: JNJ-68179280

INTERVENTIONS:
Drug: JNJ-68179280 — JNJ-68179280 will be administered as an oral capsule.
Other: Placebo — Matching placebo will be administered as an oral capsule.
  Arms: Part 1: Single Ascending Dose (SAD); Part 2: Multiple Ascending Dose (MAD)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of JNJ-68179280 compared with placebo after administration of single ascending oral doses of JNJ-68179280 administered to healthy participants (Part 1), multiple ascending oral doses of JNJ-68179280, administered to healthy participants once daily (Cohorts 1 through 4) or twice daily (Cohort 5) over 14 consecutive days (Part 2) and multiple ascending oral doses of an alternative JNJ-68179280 formulation, administered to healthy participants once daily over 14 consecutive days (Part 3 if conducted).

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening. Any abnormalities must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel (excluding liver enzymes) including hematology, blood coagulation, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Have the following pre study intervention clinical laboratory values during screening and check-in to the unit (Day -2 or Day -1): a. aspartate transaminase (AST) less than or equal to (<=) upper limit of normal (ULN), b. alanine aminotransferase (ALT) <= ULN, c. bilirubin <= ULN, d. alkaline phosphatase <= ULN, e. gamma-glutamyl transpeptidase (GGTP) <= ULN, f. albumin greater than or equal to (>=) lower limit of normal (LLN)
* A woman must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) at screening and a negative urine pregnancy test at check-in to the unit on Day -2 or Day -1
* Must be a non-smoker (not smoked for at least 6 months prior to screening) and has not used nicotine-containing products (example: nicotine patch, vaping, hookah) for 3 months prior to screening

Exclusion Criteria:

* History of liver or renal insufficiency significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* History of malignancy before screening (exceptions are squamous or basal cell carcinomas of the skin and carcinoma in situ of the cervix as long as they are considered cured with minimal risk of recurrence)
* Has an active, acute or chronic infection
* Has taken any disallowed therapies, concomitant therapy before the planned first dose of study intervention
* Has a positive urine drug screen and/or alcohol breath test during screening or on Day 2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 35 days
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs) | Up to 35 days
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to 35 days
  Number of participants with clinically significant abnormalities in vital signs (including temperature [oral or tympanic], pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Number of Participants with Clinically Significant Abnormalities in Physical Examination | Up to 35 days
  Number of participants with clinically significant abnormalities in physical examination (including general appearance, respiratory, cardiovascular, assessment through skin or oral mucosa) will be reported.
Number of Participants with Clinically Significant Abnormalities in Laboratory Safety Tests | Up to 35 days
  Number of participants with clinically significant abnormalities in laboratory safety tests (such as serum chemistry, hematology and urinalysis) will be reported.
Number of Participants with Clinically Significant Abnormalities in 12-lead Electrocardiograms (ECGs) | Up to 28 days
  Number of participants with clinically significant abnormalities in ECGs will be reported.

SECONDARY OUTCOMES:
Part 1, 2 and 3: Plasma Concentration of JNJ-68179280 | Up to 19 days
  Plasma concentration of JNJ-68179280 will be reported.
Part 1, 2 and 3: Urine Concentration of JNJ-68179280 | Up to 19 days
  Urine samples will be analyzed to determine the concentration of JNJ-68179280.
Part 1, 2 and 3: Stool Concentration of JNJ-68179280 | Up to 16 days
  Stool samples will be analyzed to determine the concentration of JNJ-68179280.
Part 1: Plasma Concentration of JNJ-68179280 Under Fasted Condition | Up to Day 6
  Plasma concentration of JNJ-68179280 under fasted condition will be reported.
Part 1: Plasma Concentration of JNJ-68179280 Under Fed Condition | Up to 13 days
  Plasma concentration of JNJ-68179280 under fed condition will be reported.
Part 1: Stool Concentration of JNJ-68179280 Under Fasted Condition | Up to Day 6
  Stool samples will be analyzed to determine the concentration of JNJ-68179280 under fasted condition.
Part 1: Stool Concentration of JNJ-68179280 Under Fed Condition | Up to 13 days
  Stool samples will be analyzed to determine the concentration of JNJ-68179280 under fed conditions.
Part 1: Number of Participants with TEAEs Under Fasted Condition | Up to 16 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Part 1: Number of Participants with TEAEs Under Fed Condition | Up to 23 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Part 1: Number of Participants with SAEs Under Fasted Condition | Up to 16 days
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 1: Number of Participants with SAEs Under Fed Condition | Up to 23 days
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 1: Number of Participants with Clinically Significant Abnormalities in Vital Signs Under Fasted Condition | Up to 16 days
  Number of participants with clinically significant abnormalities in vital signs (including temperature [oral or tympanic], pulse/heart rate, respiratory rate, and blood pressure) under fasted condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in Vital Signs Under Fed Condition | Up to 23 days
  Number of participants with clinically significant abnormalities in vital signs (including temperature [oral or tympanic], pulse/heart rate, respiratory rate, and blood pressure) under fed condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in Physical Examination Under Fasted Condition | Up to 16 days
  Number of participants with clinically significant abnormalities in physical examination (including general appearance, respiratory, cardiovascular, assessment through skin or oral mucosa) under fasted condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in Physical Examination Under Fed Condition | Up to 23 days
  Number of participants with clinically significant abnormalities in physical examination (including general appearance, respiratory, cardiovascular, assessment through skin or oral mucosa) under fed condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in Laboratory Safety Tests Under Fasted Condition | Up to 16 days
  Number of participants with clinically significant abnormalities in laboratory safety tests (such as serum chemistry, hematology and urinalysis) under fasted condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in Laboratory Safety Tests Under Fed Condition | Up to 23 days
  Number of participants with clinically significant abnormalities in laboratory safety tests (such as serum chemistry, hematology and urinalysis) under fed condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in 12-lead ECGs Under Fasted Condition | Up to 16 days
  Number of participants with clinically significant abnormalities in ECGs under fasted condition will be reported.
Part 1: Number of Participants with Clinically Significant Abnormalities in 12-lead ECGs Under Fed Condition | Up to 23 days
  Number of participants with clinically significant abnormalities in ECGs under fed condition will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency